CLINICAL TRIAL: NCT02326792
Title: Effect of Volume Training on Endurance of Trunk Extensor Muscles in Healthy Subjects: A Randomized Control Trial.
Brief Title: Effect of Volume Training on Back Endurance
Acronym: Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Collaborators: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Rubens Alexandre da Silva Jr, Titular professor, Universidade Norte do Paraná
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Unopar-Rubens-2
Record Dates: First submitted 2014-12-17; First posted 2014-12-30 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Back Pain
Keywords: Exercise; Training; Low back Pain; Physical Therapy
MeSH Terms: conditions — Back Pain; Motor Activity; Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- G1-Three sets of exercise (Experimental): G1 group - the participants will perform three sets of 15-20 repetitions of the trunk extensor exercise on a roman chair machine with the hips at 45 degrees relative to horizontal; performing trunk flexion-extension cycles for a total of 4 seconds (2 s concentric and 2 s eccentric contraction). The relative load for initial training will be placed at 20% back maximal voluntary contraction (MVC) and will be progressive during the training. The time session of training will be of 10 weeks.
  Interventions: Other: Exercise
- G2-One set of exercise (Experimental): G2 group - the participants will perform only one set of 15-20 repetitions of the trunk extensor exercise on a roman chair machine with the hips at 45 degrees relative to horizontal; performing trunk flexion-extension cycles for a total of 4 seconds (2 s concentric and 2 s eccentric contraction). The relative load for initial training will be placed at 20% back maximal voluntary contraction (MVC) and will be progressive during the training. The time session of training will be of 10 weeks.
  Interventions: Other: Exercise
- G3-Control (No Intervention): G3 group - the participants will be the control group, which not participating of exercise program in any time during the study.

INTERVENTIONS:
Other: Exercise — The groups will perform the trunk extensor exercise on a roman chair by 2 x week, for a total of 10 weeks of training (20 sessions). The load will be progressive and tested to each 14 days with regard to the number of repetition reached by the participant. The exercise is safe and will be supervised by a health sport professional.
  Arms: G1-Three sets of exercise; G2-One set of exercise

SUMMARY:
The fatigue of the trunk extensor muscles is often reported in people with the chronic low back pain (LBP). Evidences have showed that the strengthening muscular by the training of the lumbar spinal muscles is efficient to decrease the pain and disability symptoms of patients with the chronic LBP. Also, some studies have reported improve of the strength and endurance of the back muscles from of this type of training muscular. However, the exercise prescription for the trunk extensor muscles during the training is still not clear in the literature. In fact, no study has showed any differences between one and three sets of specific lumbar exercise with regard to better prescription of training in healthy subjects (e.g; preventive action) as well as in LBP subjects (e.g; intervention action).

DETAILED DESCRIPTION:
The purpose of this study is to compare an endurance trunk extensor training using one and three sets of exercise repetition on gains of strength and endurance muscular in healthy subjects.

Forty-two healthy voluntaries (from 18 to 35 years) of both the sexes will participate of this study. All participants will sign an informed consent form approved by the North of Parana University Ethics Committee for Research on Human Subjects. The sample will be randomized in three groups by the allocation from printed cards sequentially numbered in opaque envelopes: (G1, n=14) the participants will perform three sets of 15-20 repetitions of the trunk extensor exercise on a roman chair machine with the hips at 45 degrees relative to horizontal; performing trunk flexion-extension cycles for a total of 4 seconds (2 s concentric and 2 s eccentric contraction); (G2) the participants will perform only one set of 15-20 repetitions of the trunk extensor exercise on a roman chair machine with the hips at 45 degrees relative to horizontal; performing also trunk flexion-extension cycles for a total of 4 seconds (2 s concentric and 2 s eccentric); and (G3) the participants will be the control group, which not participating of any exercise program in any time during the study. A total of 10 weeks of training will be performed in the study, by 2 x week with the progression of load volume (increase the load if the total repetition of 20 is reached).

Before and after the lumbar training, all participants will be assessed by the endurance muscular (Isometric Sorensen test using time-limit, Dynamic endurance using the number of repetition, Borg fatigue perception scale and EMG surface of trunk extensor muscles by computation of median frequency fatigue estimate); and by the strength muscular (back isometric maximal voluntary contraction using a dynamometer on a roman chair). An evaluator trained will perform all testing assessment, in baseline time and after weeks of training. The evaluator will be blinded with regard the groups on assessment. Also, an exercise professional of sport will be responsible by exercise prescription to prescript the training at the Fitness center in the UNOPAR University; This professional will be also blinded to the groups.

An ANOVA two-way to compare the effects in the three groups (G1, G2, and G3) and the two times session-1: baseline and session-2: after 10 weeks); and the effects of interaction (Groups X Times) also will be tested. When necessary a Tukey post hoc analysis will be performed to localize the differences on the three groups. The effect size on each group will be calculated to determine the rate of changes from the training intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects only and not using ergogenic substances and anabolic steroids, and drugs use for increasing ot the muscular performance.
* All subjects need to be voluntaries.

Exclusion Criteria:

* Any contraindication to physical exercise performance in accord with the American College of Sports Medicine Standard Position;
* Several spinal pathologies (fractures, tumors, and inflammation), nerve root disorders (disc herniation and ,spondylolisthesis with neurological compromise, spinal stenosis, and others), several cardiorespiratory diseases, previous back surgery or pregnancy;
* Mental or physical illnesses problems that interfere with the exercise;
* Any surgery in the spine in the last 6 months;
* Upper body mass (trunk, upper limbs and head) greater than 50% of the total strength of the trunk extensor muscles from first day the data collection.
* Subjects enrolled in any exercise program outside of the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Isometric endurance (Classic Sorensen test) | 10 weeks
  To determine the improve of endurance muscular, the time-limit in seconds will be computed from modified Sorensen test executed on a roman chair. To measure the fatigue muscular, the participant would hold the unsupported trunk horizontally (Sorensen test).

SECONDARY OUTCOMES:
Number of repetitions | 10 weeks
  To determine the improve of dynamic back endurance, a second test will be performed and the number of repetitions will be computed from trunk flexion-extension cycles executed on a roman chair (2 seconds of concentric and 2 seconds of eccentric contraction; by a total of 4 seconds for each cycle).

OTHER OUTCOMES:
EMG fatigue index | 10 weeks
  The slope of median frenquency (MF) from EMG surface signals of the trunk extensor muscles (EMG fatigue estimate) will computed before and after the training during the Soresen test.
Isometric strength (maximal voluntary contractio: MVC) | 10 weeks
  All subjects will perform a maximal voluntary contraction (MVC) before and after the training, on a roman chair adaptated by a load cell to calcule the maximal strength of the back muscles at the trunk horizontal position. Three MVC will be computed and the best value will be used as outcome results.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens A DA SILVA, PhD, Study Director — Universidade Norte do Paraná

REFERENCES:
- [Background] da Silva RA, Lariviere C, Arsenault AB, Nadeau S, Plamondon A. Pelvic stabilization and semisitting position increase the specificity of back exercises. Med Sci Sports Exerc. 2009 Feb;41(2):435-43. doi: 10.1249/MSS.0b013e318188446a. PMID 19127180
- [Background] Lariviere C, Da Silva RA, Arsenault AB, Nadeau S, Plamondon A, Vadeboncoeur R. Specificity of a back muscle roman chair exercise in healthy and back pain subjects. Med Sci Sports Exerc. 2011 Jan;43(1):157-64. doi: 10.1249/MSS.0b013e3181e96388. PMID 20508534
- [Background] Verna JL, Mayer JM, Mooney V, Pierra EA, Robertson VL, Graves JE. Back extension endurance and strength: the effect of variable-angle roman chair exercise training. Spine (Phila Pa 1976). 2002 Aug 15;27(16):1772-7. doi: 10.1097/00007632-200208150-00016. PMID 12195070